CLINICAL TRIAL: NCT03406325
Title: Assessment of Mast Cell Activation Diagnostic Test in Patients With Allergic Disease
Brief Title: Mast Cell Activation Test in Allergic Disease
Status: Completed | Type: Observational
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Collaborators: Chinese University of Hong Kong (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Lee Tak Hong, Director Allergy Centre, Hong Kong Sanatorium & Hospital
Other Study IDs: REC-2017-17
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Asthma; Mastocytosis; Mast Cell Activation Syndrome; Food Allergy; Chronic Idiopathic Urticaria; Anaphylaxis; Eczema
Keywords: mast cell; allergy; genomic; biomarkers
MeSH Terms: conditions — Asthma; Mastocytosis; Mast Cell Activation Syndrome; Food Hypersensitivity; Chronic Urticaria; Anaphylaxis; Eczema; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples for mediator measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- urticaria: Patients with this condition
- asthma: Patients with this condition
- eczema: Patients with this condition
- food allergy: Patients with this condition
- anaphylaxis: Patients with this condition
- mastocytosis: Patients with this condition
- mast cell activating syndrome: Patients with this condition

SUMMARY:
Activation of mast cells in the immune system is known to cause allergic reactions sometimes with severe systemic symptoms. The investigators have recently developed a blood-based mast cell activation diagnostic test in which levels of functional activation in-vitro in primary cultured mast cells generated from the peripheral blood of single individuals can be assessed. It is the hypothesis that the test can be used to predict the potential state of in-vivo mast cell activation in any individual based on the functional activation profiles exhibited by their cultured mast cells. The investigators now wish to translate their in-vitro findings in a pilot study to disease groups where mast cell activation is expected to be high. These include highly allergic individuals; those with chronic idiopathic urticaria; those with mastocytosis; and those with the mast cell activation syndrome. Furthermore, they will use the functional genomics approach to identify gene expression biomarkers that are correlated with such diseases. The results will be compared with data that have been collected from a cohort of healthy control blood donors.

DETAILED DESCRIPTION:
The objective of this study is to assess whether patients with severe allergic diseases exhibit high levels of mast cell activation as determined by the mast cell activation diagnostic test the investigators have developed. They anticipate that patients with history of severe allergic reactions will show up as high responders in the blood-based mast cell activation diagnostic test. Moreover, using microarray analysis as the approach for gene expression studies, they anticipate further that genomics biomarkers that are correlated with the high functional activation of the in-vitro mast cells derived from these patients can be readily identified.

About 100 ml of peripheral venous blood from individual patients will be drawn into heparinized syringes and collected in a blood-collecting bag/tube containing silica. The bag/tube will be promptly processed for the generation of primary human mast cell cultures using the protocol that has previously been developed [Inflammation Research 66: 25 (2017). After culturing for 9 weeks, the resulting human mast cells will be analyzed for both their functional activity in terms of histamine release in response to the activation of high-affinity Immunoglobulin E (IgE) receptors in these cells and their gene expression profiles using microarray analysis. The in-vitro functional and genomics data will be correlated with specific diagnoses and measurements of blood prostaglandin D2 (PGD2), PGD2 metabolites, tryptase and histamine levels in blood. For mediator assays, plasma from each subject will be collected after the cluster of differentiation 34 positive (CD34+) isolation step and the samples will be aliquoted and frozen at -80 degrees centigrade for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

Any patients with the above diagnoses -

Exclusion Criteria:

Children < 18 years old; those who are unwilling or unable to donate blood; pregnant mothers.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Highly allergic individuals
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tak H Lee, Principal Investigator — Hong Kong Sanatorium and Hospital
Locations (1):
- Hong Kong Sanatorium & Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tam IYS, Ng CW, Tam SY, Lau HYA. Novel six-week protocol for generating functional human connective tissue-type (MCTC) mast cells from buffy coats. Inflamm Res. 2017 Jan;66(1):25-37. doi: 10.1007/s00011-016-0989-z. Epub 2016 Sep 15. PMID 27628164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 patients were recruited in the study. 12 were used for validation. 7 were used for patient-specific testing. Therefore, there were 1 validation group and 7 individuals' result.
Groups:
- Validation Group: Mast cell activation test employing normal donor cultured mast cells and allergic patient serum samples
- SH#1: Male patient, Total IgE: 28918KU/L; Der p2IgE: 64.4KU/L; clinical diagnosis: Eczema
- SH#2: Male patient, Total IgE: 22311KU/L; Der p2IgE: 91.24KU/L; clinical diagnosis: Eczema
- SH#3: Female patient, Total IgE: 5333KU/L; Der p2IgE: >100KU/L; clinical diagnosis: Eczema
- SH#4: Male patient, Total IgE: 4070KU/L; Der p2IgE: >100KU/L; clinical diagnosis: Eczema, Urticaria
- SH#5: Male patient, Total IgE: 379KU/L; Der p2IgE: 0.15KU/L; clinical diagnosis: Exercise-induced anaphylaxis
- SH#6: Female patient, Total IgE: 13KU/L; Der p2IgE: <0.1KU/L; clinical diagnosis: Mast cell activation syndrome
- SH#7: Male patient, Total IgE: 67KU/L; Der p2IgE: None KU/L; clinical diagnosis: Urticaria
Period: Overall Study
Arm/Group | Validation Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
Started | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: During recruitment period, no participants with asthma, food allergy, mastocytosis were recruited.
Groups:
- Total: Total of all reporting groups
Arm/Group | Validation Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7 | Total
Number analyzed (Participants) | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 11
  Male | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 7
Clinical diagnosis [Count of Participants; unit: Participants] — Clinical diagnosis of participants before Mast cell activation test
  Participants
    Eczema | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 7
    Rhinitis | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
    Urticaria | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
    Exercise-induced anaphylaxis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Mast cell activation syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Eczema and Urticaria | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mast Cell Activation Test Results for Validation Group
Description: Mast Cell Activation Test results of high/low level of house dust mite sensitivity by using normal donor cultured mast cells for validation.
Time Frame: Mast cells studied after 9 weeks in culture
Population: Mast cells were cultured from blood of normal donors to validate the (Mast Cell Activation) MAT assay. The serum samples were obtained from allergic patients with sensitivities to Der p2 and used for passive sensitization of normal donor mast cells followed by their activation by Der p2 allergen. Data were collected only from the validation group.
Measure: Count of Participants; unit: Participants
Arm/Group | Validation Group
Number analyzed (Participants) | 12
Participants
  High level of house dust mite sensitivity: number analyzed (Participants) | 8
  High level of house dust mite sensitivity: MAT positive | 6
  High level of house dust mite sensitivity: MAT negative | 2
  Low level of house dust mite sensitivity: number analyzed (Participants) | 4
  Low level of house dust mite sensitivity: MAT positive | 0
  Low level of house dust mite sensitivity: MAT negative | 4

2. Primary Outcome: Evaluation of Patient's Serum for Autoreactivity on Normal Average Responder Mast Cell Activation
Description: Patient's serum was incubated with mast cells derived from normal donors for detection of mast cell activation as evidenced by histamine release.
Time Frame: Mast cells studied after 9 weeks in culture
Population: Serum samples were obtained from 19 patients in total, of whom 12 were in the validation group. The other 7 patients were studied more extensively in the trial and their data is reported individually in this section and thereafter.
Measure: Count of Participants; unit: Participants
Groups:
- SH#1: Male patient, Total IgE: 28918 KU/L; Der p2 IgE: 64.4 KU/L; clinical diagnosis: Eczema
- SH#2: Male patient, Total IgE: 22311 KU/L; Der p2 IgE: 91.24 KU/L; clinical diagnosis: Eczema
- SH#3: Female patient, Total IgE: 5333 KU/L; Der p2 IgE: >100 KU/L; clinical diagnosis: Eczema
- SH#4: Male patient, Total IgE: 4070 KU/L; Der p2 IgE: >100 KU/L; clinical diagnosis: Eczema, Urticaria
- SH#5: Male patient, Total IgE: 379 KU/L; Der p2 IgE: 0.15 KU/L; clinical diagnosis: Exercise-induced anaphylaxis
- SH#6: Female patient, Total IgE: 13 KU/L; Der p2 IgE: <0.1 KU/L; clinical diagnosis: Mast cell activation syndrome
- SH#7: Male patient, Total IgE: 67 KU/L; Der p2 IgE: None KiloUnits (KU)/L; clinical diagnosis: Urticaria
Arm/Group | Validation Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
Number analyzed (Participants) | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage Histamine Release by Normal Average Responder Mast Cells + Patient's Serum to Assess Autoreactivity
Description: percentage of total histamine release by normal average responder mast cells that had been activated with patient's serum
Time Frame: Mast cells studied after 9 weeks in culture
Population: Mast cells derived from the validation group is reported as a group (mean +/-SD). The other 7 allergic patients were analysed and reported individually as explained earlier.
Measure: Mean (Standard Deviation); unit: percentage of histamine released
Arm/Group | Validation Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
Number analyzed (Participants) | 12 | 1 | 1 | 1 | 1 | 1 | 1 | 1
percentage of histamine released | 2.15 (0.71) | 32.1 | 3.3 | 2.8 | 3.4 | 5.1 | 3.2 | 3.8

4. Primary Outcome: Percentage Histamine Release by Patient's Mast Cells + Immunoglobulin E (IgE)/Anti-IgE
Description: percentage of total histamine release by patient's mast cells that had been activated with anti-IgE
Time Frame: Mast cells studied after 9 weeks in culture
Population: Mast cells derived from 7 allergic patients were analysed and reported individually. Patients in the validation group were not measured for this outcome and their samples were only used to validate the assay.
Measure: Number; unit: percentage of histamine release
Arm/Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
percentage of histamine release | 11.5 | 38.3 | 69.6 | 47.9 | 36.3 | 45.5 | 41.6

5. Primary Outcome: Percentage of Histamine Release by Patient's Mast Cells + Patient's Serum + Allergen
Description: Percentage of total histamine release when patient's mast cells were activated with patient's own serum and Der p2. Each patient's results are reported individually.
Time Frame: Mast cells studied after 9 weeks in culture
Population: as for outcome 4
Measure: Number; unit: percentage of histamine release
Arm/Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
percentage of histamine release | 24.5 | 54.7 | 79 | 8.4 | 0.2 | 0.2 | 0

6. Primary Outcome: Cell Yield Per 100ml Blood
Description: Cell yield of patient's mast cell culture after 9 weeks in culture as an index of cell growth and differentiation.
Time Frame: Mast cells studied after 9 weeks in culture
Population: as for outcome 4
Measure: Number; unit: Cell yield per 100ml blood
Arm/Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Cell yield per 100ml blood | 14045000 | 2895522 | 115294 | 625263 | 4867778 | 352000 | 1400000

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Validation Group | SH#1 | SH#2 | SH#3 | SH#4 | SH#5 | SH#6 | SH#7
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/12 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03406325/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03406325/ICF_001.pdf